CLINICAL TRIAL: NCT03699345
Title: Post-Market Clinical Follow-up Study to Monitor Device Performance and Outcomes of the CENTERA Transcatheter Heart Valve System
Brief Title: CENTERA PMCF: Post-Market Follow-up of the CENTERA Transcatheter Heart Valve System
Status: Completed | Type: Observational
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 2017-07
Record Dates: First submitted 2018-10-04; First posted 2018-10-09 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Aortic Valve Stenosis
Keywords: CENTERA; THV; Transcatheter Heart Valve
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Edwards CENTERA THV
  Interventions: Device: Transcatheter Aortic Valve Replacement (TAVR)

INTERVENTIONS:
Device: Transcatheter Aortic Valve Replacement (TAVR) — TAVR with the Edwards CENTERA THV System and accessories

SUMMARY:
This study will monitor device performance and safety of the Edwards CENTERA Transcatheter Heart Valve (THV) system in patients with severe, symptomatic aortic valve stenosis who are indicated for aortic valve replacement.

DETAILED DESCRIPTION:
A prospective, international, single arm, multi-center post market clinical follow-up study.

ELIGIBILITY:
Inclusion Criteria:

* Severe native valve calcific aortic stenosis
* Judged by the Heart Team to be at high or greater risk for open surgical therapy (i.e. predicted risk of surgical mortality greater than or equal to 8% at 30 days, based on the Society of Thoracic Surgeons (STS) risk score and other clinical co-morbidities unmeasured by the risk calculator).

Exclusion Criteria:

* Known hypersensitivity to Nitinol (nickel or titanium)
* Evidence of intracardiac mass, thrombus, vegetation, active infection or endocarditis
* Inability to tolerate anticoagulation/antiplatelet therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients with severe, symptomatic aortic valve stenosis who are indicated for aortic valve replacement.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-08-14 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
All-Cause Mortality | 30 days
  All-cause mortality at 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Hermann Reichenspurner, Principal Investigator — UKE Hamburg-Eppendorf - University Heart Center; Prof.Dr. Stephan Windecker, Principal Investigator — Inselspital, Klinik für Kardiologie
Locations (11):
- Aarhus University Hospital, Skejby, Aarhus, Denmark
- Clinique Pasteur Toulouse, Toulouse, France
- Germany (2):
  - Johannes Gutenberg Universitaet Mainz, Mainz
  - Deutsches Herzzentrum Muenchen (DHM), München
- Universitair Medisch Centrum Utrecht, Utrecht, Netherlands
- Spain (2):
  - Vall d'Hebron University Hospital - Barcelona, Barcelona
  - Hospital Universitario Central de Asturias, Oviedo
- United Kingdom (4):
  - Brighton and Sussex University Hospital, Brighton, East Sussex
  - Royal Victoria Hospital Belfast, Belfast
  - Queen Elisabeth Hospital Birmingham, Birmingham
  - Royal Infirmary of Edinburgh, Edinburgh

IPD SHARING:
Plan to Share IPD: No